CLINICAL TRIAL: NCT00383214
Title: A Phase III, Randomized, Double Blind, Placebo Controlled, Multi-Center Study of Epratuzumab in Patients With Active Systemic Lupus Erythematosus.
Brief Title: Study of Epratuzumab in Systemic Lupus Erythematosus (SLE)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SL0004(IMMU-103-04); EudraCT #: 2005-000706-31
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus,; antibody,; B-cell immunotherapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — epratuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epratuzumab (Active Comparator): 360 mg/m2 or 720 mg/m2 delivered by slow intravenous infusion
  Interventions: Drug: Epratuzumab
- Placebo (Placebo Comparator): Intravenous
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Epratuzumab — 360 mg/m2 or 720 mg/m2 delivered by slow intravenous infusion
  Arms: Epratuzumab
Other: Placebo — Intravenous
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Epratuzumab with standard treatments for patients with SLE.

ELIGIBILITY:
Inclusion Criteria:

* +ANA at screening
* BILAG Index B Level Activity in at least 2 body systems/organs
* Has SLE by ACR revised criteria (meets,<4 criteria)

Exclusion Criteria:

* Active Severe Lupus as defined by BILAG Index Level A in any body system or organ.
* Allergy to human antibodies or Murine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-05; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Patient response variable (complete response, partial response, non-response) evaluated at 24 weeks

SECONDARY OUTCOMES:
Proportion of patients with complete response or partial response;
Individual BILAG assessments;
Physician and patient assessment scores;
Time-to treatment failure;
Successful steroid reduction by weeks 20 and 24;
Maintenance of steroid reduction at 24 and 48 weeks;
Monitor the plasma concentration and immunogenicity profile of epratuzumab in patients with Lupus;
Assess epratuzumab on Health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Anna Barry, Study Director — UCB Pharma
Locations (60):
- United States (25):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Los Angeles, California
  - Upland, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Farmington, Connecticut
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Chicago, Illinois
  - Baltimore, Maryland
  - New York, New York
  - Plainview, New York
  - Rochester, New York
  - Syracuse, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Gallipolis, Ohio
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - Arlington, Virginia
  - Edmonds, Washington
- Belgium (2):
  - Brussels
  - Liège
- Brazil (5):
  - Rio de Janeiro, Rio de Janeiro
  - Goiânia
  - Rio de Janeiro
  - São Paulo
  - Sorocaba
- Canada (2):
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
- Czechia (3):
  - Hradec Králové
  - Olomouc
  - Prague
- France (2):
  - Paris
  - Toulouse
- Germany (4):
  - Erlangen
  - Heidelberg
  - Mannheim
  - München
- Italy (2):
  - Ancona
  - Brescia
- Netherlands (3):
  - Amsterdam
  - Groningen
  - Leiden
- Spain (5):
  - Barcelona
  - Madrid
  - San Cristóbal de La Laguna
  - Santander
  - Seville
- United Kingdom (7):
  - Leeds, West Yorkshire
  - Birmingham
  - London
  - Manchester
  - Newcastle upon Tyne
  - Sheffield
  - United Kingdom

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069